CLINICAL TRIAL: NCT04774367
Title: Evaluation of the Reliability of the Determination of MisMatch Repair Deficiency Status by Endoscopic Biopsies in Oesophagus and Gastric Adenocarcinoma.
Acronym: BIOPSYGAST MMR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP180152
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Gastro-oesophageal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps (Other)
  Interventions: Device: Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps
- Order of forceps : First large capacity biopsy forceps and second standard biopsy forceps (Other)
  Interventions: Device: Order of forceps : First large capacity biopsy forceps and second standard biopsy forceps

INTERVENTIONS:
Device: Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps — Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps
  Arms: Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps
Device: Order of forceps : First large capacity biopsy forceps and second standard biopsy forceps — Order of forceps : First standard biopsy forceps and second large capacity biopsy forceps
  Arms: Order of forceps : First large capacity biopsy forceps and second standard biopsy forceps

SUMMARY:
Gastro-esophageal adenocarcinoma is one of the most common cancer in the world and the fourth most common cancer in France with more than 6,000 cases per year. For non-metastatic patients, a preoperative chemotherapy is recommended.

As colorectal adenocarcinomas, gastroesophageal cancers (OGC) could be caused by a failure of DNA repair related to the loss of expression of one of the DNA repair proteins (MLH1, MSH2, PMS2, MSH6) (deficient MMR (dMMR)). The prevalence of tumors with dMMR is evaluated at 14% (Choi et al, 2014; Kim et al, 2015). This proportion reaches 25% among patients over 70 years old. Evidence suggests that patients with dMMR tumors do not benefit from neoadjuvant chemotherapy (Smyth et al, 2017), which may even have a negative impact, especially in elderly patients, and which should be discussed in this particular situation. The decision of neo-adjuvant chemotherapy must be taken very quickly after the endoscopic diagnosis.

The investigators will evaluate the diagnostic performance of the determination of dMMR status by endoscopic biopsies of OGC.

Moreover, there is no clear recommendation for the determination of dMMR status in OGC especially regarding the size of the forceps to use to ensure the quality of samples and the best molecular techniques for dMMR status determination.

Methods In this prospective study, the investigators will include patients who will benefit from an upper endoscopy within 5 French hospital centers (Saint-Louis, Lariboisière, Beaujon, Bichat and Avicenne) linked to the NORDICAP network. If a suspect lesion of OGC is discovered during the gastroscopy, the endoscopist will perform at least 8 endoscopic biopsies, according to the recommendations, and by the mean of 2 kinds of forceps: standard biopsy forceps and a large capacity biopsy forceps. The clinical and follow-up data will be prospectively collected and will include demographics data, cancer stage, lymph node invasion, treatment history, recurrence and survival data. The investigators will assess MSI status by genotyping and MMR proteins expression by immunochemistry (IHC), performed, for each patient, on both biopsies and surgical tumor samples.

Expected results This study will allow us to compare diagnostic performance of endoscopic biopsies to surgical samples for the assessment of dMMR status. Likewise, the investigators will compare the diagnostic performance of the two kinds of endoscopic forceps and of IHC and genotyping for the determination of dMMR phenotype. It will enable us to establish recommendations for the benefit of gastro-enterologists and pathologists.

ELIGIBILITY:
Eligible criteria :

* Patient having endoscopic oesogastroduodenal endoscopy for suspicion of oesogastro-duodenal adenocarcinoma.
* Benefiting from the social security system

Inclusion Criteria:

* Patient having endoscopy biopsies in front of a suspicious lesion suggestive of gastroesophageal adenocarcinoma

Exclusion Criteria:

* Minor patient (<18 years old)
* known pregnancy
* Major patient under tutorship or curatorship
* Contraindication to gastric biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (Se) of the determination of the dMMR status by the endoscopic biopsies performed at the time of the initial high endoscopy | at inclusion
  The sensitivity will be evaluated by comparing the endocospic result with that obtained by the analysis of the specimen considered as the reference examination.
Specificity (Spe) of the determination of the dMMR status by the endoscopic biopsies performed at the time of the initial high endoscopy | at inclusion
  The specificity will be evaluated by comparing the endocospic result with that obtained by the analysis of the specimen considered as the reference examination.

SECONDARY OUTCOMES:
Positive likelihood ratios | at inclusion
Negative likelihood ratios | at inclusion
Sensitivity of dMMR status diagnosis according to the forceps (standard and large capacity biopsy forceps ) | at inclusion
Specificity of dMMR status diagnosis according to the forceps (standard and large capacity biopsy forceps ) | at inclusion
Sensitivity of dMMR status diagnosis according to the techniques (immunohistochemistry and PCR) | at inclusion
Specificity of dMMR status diagnosis according to the techniques (immunohistochemistry and PCR) | at inclusion
Sensitivity of the diagnosis of MR status according to the location on the biopsies (esophagus, gastroesophageal junction, fundus, antrum) | at inclusion
Specificityof the diagnosis of MR status according to the location on the biopsies (esophagus, gastroesophageal junction, fundus, antrum) | at inclusion
Sensitivity of dMMR status diagnosis according to the number of techniques used (two techniques or one technique) | at inclusion
Specificity of dMMR status diagnosis according to the number of techniques used (two techniques or one technique) | at inclusion
Overall survival | up to 36 months
Survival without recurrence | up to 36 months

IPD SHARING:
Plan to Share IPD: Undecided